CLINICAL TRIAL: NCT03532698
Title: Prospective Observational Trial to Evaluate the Efficacy of the Combination of Osimertinib and Aspirin in Patients With Disease Progression to 3st Generation Epidermal Growth Factor Receptor-tyrosine Kinase Inhibitor（EGFR-TKI） Osimertinib
Brief Title: Combination of Osimertinib and Aspirin to Treat Osimertinib Resistance Non-small Cell Lung Cancer ( NSCLC)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Yong He, Daping Hospital and the Research Institute of Surgery of the Third Military Medical, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Other Study IDs: COAST 2
Record Dates: First submitted 2018-04-24; First posted 2018-05-22 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Non-Small Cell Lung Cancer Stage IIIB; Non-small Cell Lung Cancer Stage IV; EGFR T790M
Keywords: lung cancer; Aspirin; Osimertinib; EGFR-TKI; resistance
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Aspirin; osimertinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- osimertinib and aspirin: Osimertinib and Aspirin starting at a dose of 80 mg and 100mg once a day, orally with meals. Aspirin treatment will be initiated one week before beginning TKI therapy, if possible, but TKI therapy will not be delayed for Aspirin loading. Drug: Osimertinib and Aspirin will be administered once every day. If subject has complete response, partial response, stable disease, or unacceptable toxicity.
  Interventions: Drug: Aspirin; Drug: Osimertinib
- osimertinib: Osimertinib starting at a dose of 80 mg once a day, orally with meals. Drug: Osimertinib will be administered once every day. If subject has complete response, partial response, stable disease, or unacceptable toxicity.
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: Aspirin — Aspirin, also known as acetylsalicylic acid (ASA), is a very safe medication used to treat pain, fever, or inflammation.
  Other Names: ASP
  Groups: osimertinib and aspirin
Drug: Osimertinib — Osimertinib, also known as azd9291, is a 3rd-generation EGFR-TKI used to treat NSCLC patients with resistance to 1st generation EGFR-TKI due to T790M mutation. It has been approved in clinical applications by the FDA in 2015.
  Other Names: OSI

SUMMARY:
The third generation epidermal growth gactor receptor-tyrosine Kinase Inhibitor（EGFR-TKI） osimertinib has obvious curative effect for EGFR sensitive mutation and T790M mutation(PMID 27959700), but acquired drug resistance will occur. Previous studies show that apoptosis escape can lead to EGFR-TKI resistance.Osimertinib resistant cells show abnormal activation of PI3K/AKT/BIM activation(PMID 28765329). The classical drug aspirin can effectively decrease AKT phosphorylation and activate of BIM(PMID 28881293).So Investigators speculate that aspirin may decrease the PI3K/AKT/BIM signaling pathways, then promote osimertinib resistant cells apoptosis. The current study aims to evaluate the combination of aspirin and osimertinib in patients with EGFR/T790M mutations.

DETAILED DESCRIPTION:
Reversible small-molecule EGF receptor tyrosine kinase inhibitors (EGFR-TKI) have shown dramatic therapeutic efficacy in non-small cell lung cancer (NSCLC) patients with EGFR-activating mutations, and have been recommended as the standard first-line therapy in these patients. However, despite excellent initial clinical responses, nearly all patients eventually develop drug resistance after a median period of about 10 months(PMID 26497205). Osimertinib is a 3rd-generation EGFR-TKI used to treat NSCLC patients with resistance to 1st generation EGFR-TKI due to T790M mutation. But Osimertinib also face the problem of acquired drug-resistance(PMID 27959700). Thus, innovative treatment strategies are urgently needed to overcome therapeutic resistance to Osimertinib to improve the survival of patients with NSCLC.

Molecular mechanisms underlying acquired Osimertinib resistance are still not fully understood. Previous study showed that one principal mechanism accounting for majority of acquired resistance to Osimertinib in lung cancer is mediated by an exon 20 C797S mutation etc(PMID 29596911). More molecular mechanisms are still to be found. Apoptosis is a process of programmed cell death that occurs in multicellular organisms. Biochemical events lead to characteristic cell changes (morphology) and death. These changes include blebbing, cell shrinkage, nuclear fragmentation, chromatin condensation, chromosomal DNA fragmentation, and global mRNA decay. Apoptosis has been found to be related to drug resistance to 1st generation EGFR-TKI(PMID 29731879). The investigators previous found apoptosis is also related to Osimertinib resistance(PMID 28765329). Therefore, promoting apoptosis may be an effective way to improve the response to Osimertinib treatment.

Investigators' group has focused on lung cancer targeted therapy for several years. Previously, investigators have reported that metformin in combination with 1st generation EGFR-TKI could enhance the effect of TKI (PMID 24644001). Therefore, investigators further asked whether the drug combination approach could overcome osimertinib resistance. Aspirin is a widely used and well-tolerated drug for Kawasaki disease, pericarditis, and rheumatic and has arisen keen interest as a potential anticancer agent ever since the report of the clinical evidence that the cancer risk and mortality are reduced in Colon cancer. Aspirin exerts remarkable antitumor properties in tumor cells and mouse models. It strongly inhibited the growth of lung cancer cells, and its combination with TKI agents, including Sorafenib (PMID: 28857200), significantly suppressed RAS-mutant cancers growth and prolonged remission in a xenograft model. Interestingly, Aspirin exposure significantly promoted the apoptosis suggesting that aspirin may overcome Osimertinib resistance by promoting the apoptosis.

Here, investigators'group observed that in clinic, several patients who took osimertinib and aspirin together have shown excellent effect.Investigators therefore conduct this clinical trial to observe whether the combination of Aspirin and Osimertinib could enhance efficacy of Osimertinib in lung cancer patients resistant to 1st generation EGFR-TKI with T790M.

ELIGIBILITY:
Inclusion Criteria:

•Patients must have Histologically or cytologically confirmed non small cell carcinoma of the lung who harbors EGFR-mutation and are previously disease progression to 3st generation EGFR-TKI Osimertinib.

Patient must have measurable stage IV disease (includes M1a, M1b stages or recurrent disease) (according to the 7th edition of the tumor node metastasis (TNM) classification system). However, patients with T4NX disease (stage III B) with nodule(s) in ipsilateral lung lobe are not eligible, because such patients were not included in historical controls.

* Patients be age >18 years and < 75 years.
* Patients must have a Life Expectancy of greater than 12 weeks.
* Patients must have an electrocorticography (ECOG) performance status 0 or 1 (Karnofsky > 70).
* Patients must have normal organ and marrow function as defined below, within one week prior to randomization: absolute neutrophil count >1,500/mL platelets > 100,000/mL total bilirubin: within normal institutional limits AST(SGOT)/ALT(SGPT) < 2.5 X institutional upper limit of normal creatinine < 1.5 X institutional upper limit of normal urine dipstick for proteinuria of < less than 1+. If urine dipstick is > 1+ then a 24 hour urine for protein must demonstrate < 500 mg of protein in 24 hours to allow participation in the study.

Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

* Patients must have an international normalized ratio (INR) < 1.5 and a partial thromboplastin time (PTT) no greater than upper limits of normal within 1 week prior to randomization.
* Patients with a history of hypertension must be well-controlled (<150 systolic/<100 diastolic) on a stable regimen of anti-hypertensive therapy.
* Patients must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection,symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia,gastric ulcer,hemophilia,thrombopenia,active hemorrhage,podagra,kidney failure or psychiatric illness/social situation that would limit compliance with study requirements.
* Patients receiving chronic daily treatment with aspirin (> 325 mg/day) or nonsteroidal anti-inflammatory agents known to inhibit platelet function. Treatment with dipyridamole (Persantine), ticlopidine (Ticlid),clopidogrel (Plavix) and/or cilostazol (Pletal)is also not allowed.
* Patients receiving therapeutic anticoagulation. Prophylactic anticoagulation of venous access devices is allowed provided Section 3.10 is met. Caution should be taken on treating patients with low dose heparin or low molecular weight heparin for DVT prophylaxis during treatment with bevacizumab as there may be an increased risk of bleeding.
* Prior use of chemotherapy.
* Patients receiving immunotherapy, hormonal-therapy and or radiotherapy within 2 weeks prior to entering the study. Note: Those who have not recovered from adverse events due to these agents administered will be considered ineligible.
* Patients receiving any other investigational agents.
* Patients with uncontrolled brain metastasis. Note: Patients with brain metastases must have stable neurologic status following local therapy (surgery or radiation) for at least 2 weeks, and must be without neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to Osimertinib and Aspirin or other agents used in the study are excluded.
* Women that are pregnant or breastfeeding Note: Pregnant women are excluded from this study because the agents used in this study may be teratogenic to a fetus. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with paclitaxel, breastfeeding women are also excluded from this study.
* Patients that are HIV-positive on combination antiretroviral therapy due to the potential for lethal infections when treated with marrow-suppressive therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must have Histologically or cytologically confirmed non small cell carcinoma of the lung who harbors EGFR-mutation and are previously disease progression to 3st generation EGFR-TKI Osimertinib.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) according to resist 1.1 | 2years
  To evaluate the response to therapy and Objective Response Rate of the combination of Osimertinib and Aspirin in patients who has metastatic pulmonary adenocarcinoma disease progression to 3st generation EGFR-TKI Osimertinib.

SECONDARY OUTCOMES:
disease control rate(DCR) according to resist 1.1 | 2years
  To evaluate the response to therapy and disease control rate of the combination of Osimertinib and Aspirin in patients who has metastatic pulmonary adenocarcinoma disease progression to 3st generation EGFR-TKI Osimertinib.
Time to progression(TTP) according to resist 1.1 | 2years
  To evaluate the response to therapy and Time to progression of the combination of Osimertinib and Aspirin in patients who has metastatic pulmonary adenocarcinoma disease progression to 3st generation EGFR-TKI Osimertinib.
duration of Response(DOR) according to resist 1.1 | 2years
  To evaluate the response to therapy and duration of Response of the combination of Osimertinib and Aspirin in patients who has metastatic pulmonary adenocarcinoma disease progression to 3st generation EGFR-TKI Osimertinib.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shi P, Oh YT, Deng L, Zhang G, Qian G, Zhang S, Ren H, Wu G, Legendre B Jr, Anderson E, Ramalingam SS, Owonikoko TK, Chen M, Sun SY. Overcoming Acquired Resistance to AZD9291, A Third-Generation EGFR Inhibitor, through Modulation of MEK/ERK-Dependent Bim and Mcl-1 Degradation. Clin Cancer Res. 2017 Nov 1;23(21):6567-6579. doi: 10.1158/1078-0432.CCR-17-1574. Epub 2017 Aug 1. PMID 28765329
- [Background] Ma J, Cai Z, Wei H, Liu X, Zhao Q, Zhang T. The anti-tumor effect of aspirin: What we know and what we expect. Biomed Pharmacother. 2017 Nov;95:656-661. doi: 10.1016/j.biopha.2017.08.085. Epub 2017 Sep 4. PMID 28881293
- [Background] Li L, Han R, Xiao H, Lin C, Wang Y, Liu H, Li K, Chen H, Sun F, Yang Z, Jiang J, He Y. Metformin sensitizes EGFR-TKI-resistant human lung cancer cells in vitro and in vivo through inhibition of IL-6 signaling and EMT reversal. Clin Cancer Res. 2014 May 15;20(10):2714-26. doi: 10.1158/1078-0432.CCR-13-2613. Epub 2014 Mar 18. PMID 24644001
- [Background] Li S, Dai W, Mo W, Li J, Feng J, Wu L, Liu T, Yu Q, Xu S, Wang W, Lu X, Zhang Q, Chen K, Xia Y, Lu J, Zhou Y, Fan X, Xu L, Guo C. By inhibiting PFKFB3, aspirin overcomes sorafenib resistance in hepatocellular carcinoma. Int J Cancer. 2017 Dec 15;141(12):2571-2584. doi: 10.1002/ijc.31022. Epub 2017 Sep 14. PMID 28857200
- [Background] Minari R, Bordi P, La Monica S, Squadrilli A, Leonetti A, Bottarelli L, Azzoni C, Lagrasta CAM, Gnetti L, Campanini N, Petronini PG, Alfieri R, Tiseo M. Concurrent Acquired BRAF V600E Mutation and MET Amplification as Resistance Mechanism of First-Line Osimertinib Treatment in a Patient with EGFR-Mutated NSCLC. J Thorac Oncol. 2018 Jun;13(6):e89-e91. doi: 10.1016/j.jtho.2018.03.013. Epub 2018 Mar 27. No abstract available. PMID 29596911
- [Result] Mok TS, Wu Y-L, Ahn M-J, Garassino MC, Kim HR, Ramalingam SS, Shepherd FA, He Y, Akamatsu H, Theelen WS, Lee CK, Sebastian M, Templeton A, Mann H, Marotti M, Ghiorghiu S, Papadimitrakopoulou VA; AURA3 Investigators. Osimertinib or Platinum-Pemetrexed in EGFR T790M-Positive Lung Cancer. N Engl J Med. 2017 Feb 16;376(7):629-640. doi: 10.1056/NEJMoa1612674. Epub 2016 Dec 6. PMID 27959700